CLINICAL TRIAL: NCT02938442
Title: A Combined Phase i/II Efficacy Study of a Carbohydrate Mimotope-based Vaccine With MONTANIDE™ ISA 51 VG STERILE Combined With Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Brief Title: Vaccination of Triple Negative Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206010
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-06

CONDITIONS: Triple Negative Breast Cancer; Breast Neoplasms
Keywords: clinical stage I, II or III; TNBC; ER positive; PR positive; HER2 positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy Only Arm (Active Comparator): Subjects randomized to the control arm will receive SoC neoadjuvant chemotherapy starting on week 1. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- Chemo+Vaccine Arm (Experimental): Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Interventions: Biological: P10s-PADRE with MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Biological: P10s-PADRE with MONTANIDE™ ISA 51 VG — Subjects randomized to the control arm will receive SoC neoadjuvant chemotherapy starting on week 1. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Other Names: P10s-PADRE/ MONTANIDE™ ISA 51 VG
  Arms: Chemo+Vaccine Arm
Drug: Doxorubicin — Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
Drug: Cyclophosphamide — Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
Drug: Paclitaxel — Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.

SUMMARY:
The purpose of this study is to evaluate a new investigational cancer vaccine, P10s-PADRE in combination with standard neoadjuvant chemotherapy and surgery in patients with clinical stage I, II or III triple negative breast cancer (TNBC). This study will compare the vaccine plus standard neoadjuvant chemotherapy and surgery to standard neoadjuvant chemotherapy and surgery alone.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an investigational agent, P10s-PADRE, a peptide mimotope-based vaccine, in combination with standard neoadjuvant chemotherapy in patients with clinical stage I, II or III estrogen-receptor (ER) negative, progesterone receptor (PR) negative and HER2-negative (= triple negative - TN) breast cancer. P10s-PADRE will be administered with MONTANIDE™ ISA 51 VG as adjuvant. Human breast cancers that express Tumor Associated Carbohydrate Antigens (TACAs) can be immunogenic, and enhancing the anti-TACA antibodies and immune effector function already present may augment the cytotoxic effects of standard therapies.

A randomized two-arm, open-label, multi-center phase I/II trial is designed with the goal being to evaluate the efficacy of combining vaccination of the P10s-PADRE formulation with neoadjuvant chemotherapy. Patients will be randomly assigned in a 2:1 ratio to standard chemotherapy plus P10s-PADRE or to standard chemotherapy alone. Efficacy will be based on the rate of pathologic Complete Response (pCR) observed among TN breast-cancer patients treated with the combination as compared with the group of patients who receive standard chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Females of all races with biopsy-proven clinical stage I, II, or III TNBC (ER-negative, PR-negative and HER2-negative) who will undergo SoC neoadjuvant treatment
* Age 18 years and older
* ECOG Performance Status 0 or 1
* White blood cell (WBC) count ≥ 3,000/mm3 within 3 weeks prior to registration
* Platelet count ≥ 100,000/mm3 within 3 weeks prior to registration
* Bilirubin ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration
* Serum glutamic-oxaloacetic transaminase (SGOT) or aspartate aminotransferase test (AST) ≤ 2 x IUL of normal obtained within 3 weeks prior to registration
* Serum glutamic-pyruvic transaminase (SGPT) or alanine aminotransferase test (ALT) ≤ 2 x IUL of normal obtained within 3 weeks prior to registration
* Serum creatinine ≤ 1.8 mg/dl obtained within 3 weeks prior to registration
* Must sign an informed consent document approved by the UAMS IRB

Exclusion Criteria:

* ER-positive, PR-positive, HER2-positive, inflammatory, metastatic, stage IV or recurrent breast cancer.
* Active infection requiring treatment with antibiotics.
* Existing diagnosis or history of organic brain syndrome that might preclude participation in the full protocol.
* Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol.
* Other current malignancies. Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.
* Active autoimmune disorders or conditions of immunosuppression; Existing diagnosis or history of autoimmune disorders or conditions of immunosuppression that have been in remission for less than 6 months.
* Treatment with corticosteroids, including oral steroids (i.e. prednisone, dexamethasone [except when used as an antiemetic in SoC therapy]), continuous use of topical steroid creams or ointments or any steroid-containing inhalers. Subjects who discontinue the use of these classes of medication for at least 6 weeks prior to registration are eligible if, in the judgment of the treating physician, the subject is not likely to require these classes of drugs during the treatment period. Replacement doses of steroids for subjects with adrenal insufficiency are allowed.
* Pregnancy or breastfeeding (due to the unknown effects of peptide/mimotope vaccines on a fetus or infant). Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to starting week 1 and must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 18 months after completing or discontinuing treatment. Accepted methods of contraception include oral contraceptives, barrier methods, IUDs, and abstinence.
* Any other significant medical or psychiatric conditions, which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen.
* Enrollment in any other clinical trial using investigational drug products or devices prior to first post-surgery study lab (Week 46 visit). Concurrent enrollment in observational studies is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu Malapati, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Only: Subjects randomized to the control arm will receive SoC neoadjuvant chemotherapy starting on week 1. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Doxorubicin + Cyclophosphamide + Paclitaxel: Eligible subjects will be enrolled and receive standard neoadjuvant chemotherapy alone
- Chemo+Vaccine: Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  P10s-PADRE with MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Paclitaxel: Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period in combination with standard neoadjuvant chemotherapy.
Period: Overall Study
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Started | 5 | 11
Completed | 3 | 8
Not Completed | 2 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were randomized to the control arm, which would receive SoC neoadjuvant chemotherapy or the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Only | Chemo+Vaccine | Total
Number analyzed (Participants) | 5 | 11 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.91) | 56.55 (11.26) | 56.5 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Adverse Events
Description: A Safety/Tolerability Event is defined as the occurrence of one of the following:
  * A Serious Adverse Event, OR
  * A non-Serious Adverse Event of Grade = 3, 4, or 5, OR
  * A non-Serious Adverse Event of Grade = 2 whose Relationship to P10s-PADRE Vaccine was classified as Definite, Probable, or Possible
Time Frame: From the start of treatment to the time of definitive surgery (4-8 weeks after chemo); from Week 0 to Week 20-23
Measure: Number; unit: Total events
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Total events | 8 | 81

2. Primary Outcome: Pathologic Complete Response (pCR)
Description: A tumor-response call of either ypT0N0 or ypTisN0 determined through surgical staging after neoadjuvant therapy. The staging system used to determine the tumor-response call is the AJCC Staging System described in a 2014 FDA Guidance for Industry.
  • A tumor-response call of "pyT0N0" is also equated with pCR in the published literature.
Time Frame: During and/or Immediately After Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Participants
  Pathologic Complete Response (pCR) | 1 | 2
  No Pathologic Complete Response (pCR) | 4 | 9

3. Primary Outcome: Pathological Tumor Size
Description: Tumor size at surgery/pathology report
Time Frame: Surgery
Population: For 2 participants, there was no data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 9
centimeters | 3.52 (5.65) | 0.98 (0.85)

4. Primary Outcome: Pathological Node Status: Number of Positive Lymph Nodes
Description: Number of positive lymph nodes found out of dissected lymph nodes
Time Frame: Surgery
Population: For 3 participants, there were no data.
Measure: Mean (Standard Deviation); unit: lymph node
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 8
lymph node | 6.6 (14.76) | 1.5 (3.46)

5. Primary Outcome: Pathological Node Status: Number of Dissected Lymph Nodes
Description: Number of dissected lymph nodes at surgery for study participants
Time Frame: Surgery
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities.
Measure: Mean (Standard Deviation); unit: lymph node
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
lymph node | 10.2 (14.06) | 6.91 (5.74)

6. Primary Outcome: Tumor Response
Description: Participants had their tumors surgically removed and pathologically staged using the AJCC Staging criteria. The main method of pathologic staging for breast cancer is the TNM system which stands for (Tumor size, lymph Node status and Metastases). "yp" prior to TN means the tissue was staged after neoadjuvant therapy. The larger the number after "T" means the larger the size, and the larger the number after "N" means the number of affected nearby lymph nodes. Therefore, tumor gradings with T3Nx are worse than those with T0Nx. The two categories "pyT0N0" and "ypT0N0" are both considered to be synonymous with pCR in the published literature.
Time Frame: Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Participants
  mypT1aN | 0 | 1
  mypT1ap | 0 | 1
  mypT1b | 0 | 1
  pyT0N0 | 0 | 1
  ypT0N0 | 1 | 1
  ypT0N3a | 0 | 1
  ypT0pN1 | 0 | 1
  ypT1aN0 | 1 | 0
  ypT1cN0 | 1 | 0
  ypT1cN1 | 0 | 1
  ypT1cNX | 0 | 1
  ypT1pN0 | 0 | 1
  ypT2N0 | 1 | 1
  ypT3Na | 1 | 0

7. Secondary Outcome: Fold Increase in P10s-MAP-Reactive Immunoglobulin Titers
Description: The anti-P10s binding level was measured via ELISA method after incubation with a subject's serum samples. The endpoint titer was determined for each serum sample, and then fold change in endpoint titer in post-treatment weeks compared to pre-treatment week (Week 1) were calculated.
Time Frame: Weeks 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities.
Measure: Mean (Standard Deviation); unit: fold change in serum titer
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
fold change in serum titer
  Week 7 | 1 (0) | 2.27 (2.83)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 3 (4.80)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 1.73 (2.1)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 1.36 (0.92)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 1.55 (1.21)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 1 (0) | 5.4 (9.45)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 6.25 (10.69)

8. Secondary Outcome: Frequencies of NK Cells - CD16
Description: Using flow cytometry, the frequencies of NK cells were determined for samples collected from multiple timepoints from Week 1 to Week 70. Values were averaged for the percent of CD16+NK cells.
Time Frame: Week 1, 7, 10, 15, 18, 23, 46, 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of NK Cells
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of NK Cells
  Week 1 | 76.89 (39.81) | 90.57 (4.87)
  Week 7 | 66.72 (32.41) | 87.36 (5.84)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 69.96 (15.09)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 83.38 (7.82)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 87.79 (6.7)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 80.9 (5)
  Week 46: number analyzed (Participants) | 3 | 11
  Week 46 | 94.2 (2.63) | 82.91 (9.51)
  Week 70: number analyzed (Participants) | 0 | 11
  Week 70 |  | 96.64 (6.92)

9. Secondary Outcome: Frequencies of NK Cells - CD69
Description: Using flow cytometry, the frequencies of NK cells were determined for samples collected from multiple timepoints from Week 1 to Week 70. Values were averaged for the percent of CD69+NK cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Week 46 and Week 70, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of NK cells
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of NK cells
  Week 1 | 5.19 (2.06) | 7.89 (5.98)
  Week 7 | 3.64 (1.71) | 13.54 (5.28)
  week 10: number analyzed (Participants) | 0 | 11
  week 10 |  | 5.98 (2.49)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 15.73 (27.88)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 9.52 (7.28)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 11.21 (8.7)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 2.93 (1.21) | 6.14 (3.35)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 3.98 (1.97)

10. Secondary Outcome: Frequencies of NK Cells - NKp46
Description: Using flow cytometry, the frequencies of NK cells were determined for samples collected from multiple timepoints from Week 1 to Week 70. Values were averaged for the percent of NKp46+NK cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 1, 10, 25, 46 and 70, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of NK cells
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of NK cells
  Week 1: number analyzed (Participants) | 5 | 10
  Week 1 | 87.98 (13.41) | 77.98 (29.16)
  Week 7 | 73.64 (25.66) | 83.36 (16.84)
  Week 10: number analyzed (Participants) | 0 | 10
  Week 10 |  | 70.35 (27.32)
  Week 15: number analyzed (Participants) | 0 | 10
  Week 15 |  | 87.77 (11.01)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 90.15 (11.37)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 82.19 (28)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 77.13 (32.39) | 86.84 (10.25)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 90.31 (4.95)

11. Secondary Outcome: Frequencies of NK Cells - NKG2D
Description: Using flow cytometry, the frequencies of NK cells were determined for samples collected from multiple timepoints from Week 1 to Week 70. Values were averaged for the percent of NKG2D+NK cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 1, 46 and 70, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of NK cells
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of NK cells
  Week 1: number analyzed (Participants) | 5 | 10
  Week 1 | 90.88 (6.67) | 93.74 (4.13)
  Week 7 | 81.76 (6.54) | 89.26 (6.24)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 78.34 (15.83)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 91.66 (6.93)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 91.04 (4.94)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 91.91 (6.48)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 86.93 (8.56) | 89.33 (5.97)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 91.46 (5.32)

12. Secondary Outcome: Frequencies of T Cells - CD3+/CD4+
Description: Using flow cytometry, the frequencies of CD3+/CD4+ T cells were determined for samples collected from multiple timepoints from Week 1 to Week 46. Values were averaged for the percent of CD4 T cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, and 46
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 1,7, and 23, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of T cell
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of T cell
  Week 1: number analyzed (Participants) | 5 | 10
  Week 1 | 58.9 (16.38) | 54.64 (11.64)
  Week 7: number analyzed (Participants) | 5 | 9
  Week 7 | 45.92 (18.34) | 59.89 (10.91)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 46.59 (12.37)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 47.38 (11.60)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 48.57 (10.19)
  Week 23: number analyzed (Participants) | 0 | 9
  Week 23 |  | 43.97 (14.07)
  Week 46: number analyzed (Participants) | 3 | 11
  Week 46 | 39.83 (5.1) | 43.66 (13.72)

13. Secondary Outcome: Frequencies of T Cells - CD3+/CD8+
Description: Using flow cytometry, the frequencies of CD3+/CD8+ T cells were determined for samples collected from multiple timepoints from Week 1 to Week 46. Values were averaged for the percent of CD8 T cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, and 46
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 1, 7, 15, and 18, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of T cell
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of T cell
  Week 1: number analyzed (Participants) | 5 | 9
  Week 1 | 33.68 (12.88) | 35.62 (11.78)
  Week 7: number analyzed (Participants) | 5 | 10
  Week 7 | 46.46 (15.78) | 34.95 (13.5)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 39.90 (13.77)
  Week 15: number analyzed (Participants) | 0 | 10
  Week 15 |  | 44.95 (9.22)
  Week 18: number analyzed (Participants) | 0 | 10
  Week 18 |  | 42.6 (9.24)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 46.84 (15.6)
  Week 46: number analyzed (Participants) | 3 | 11
  Week 46 | 53.03 (3.85) | 45.99 (10.33)

14. Secondary Outcome: Frequencies of Cells - CD69+/CD3+
Description: Using flow cytometry, the frequencies of CD69+/CD3+ cells were determined for samples collected from multiple timepoints from Week 1 to Week 70. Values were averaged for the percent of CD69 T cells.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 46 and 70, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of T cell
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
percentage of T cell
  Week 1 | 3.17 (2.21) | 4.57 (2.55)
  Week 7 | 2.52 (1.54) | 9.86 (8.33)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 4.61 (2.87)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 14.38 (27.03)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 8.17 (6.23)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 10.25 (7.74)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 2.55 (0.92) | 9 (14.51)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 4.02 (2)

15. Secondary Outcome: Frequencies of Circulating Regulatory T Cells (Tregs)
Description: Peripheral blood mononuclear cells (PBMCs) were isolated from samples collected from multiple timepoints from Week 1 to Week 46. Using flow cytometry, the frequencies of Tregs (CD4, CD25 and CD127) were analyzed for separately, and then summed. The units are reported in CD4+CD25+CD127 low/- percentage because CD127 is a recently discovered antigen associated with Tregs that is weakly expressed on Tregs, while the self-activated memory T cell CD127 is strongly expressed; therefore, CD4+CD25+CD127 low/- is used to represent Tregs now.
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm, Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm, Weeks 1, 7, 10, 15, 46 and 70, participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: percentage of Tcell CD4+CD25+CD127low/-
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 3 | 11
percentage of Tcell CD4+CD25+CD127low/-
  Week 1: number analyzed (Participants) | 3 | 10
  Week 1 | 9.68 (3.83) | 9.04 (3.37)
  Week 7: number analyzed (Participants) | 3 | 10
  Week 7 | 10.8 (4.59) | 5.27 (1.98)
  Week 10: number analyzed (Participants) | 0 | 10
  Week 10 |  | 8.26 (2.58)
  Week 15: number analyzed (Participants) | 0 | 10
  Week 15 |  | 8.82 (3.97)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 5.75 (2.08)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 8.48 (1.7) | 12.88 (6.25)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 9.37 (2.25)

16. Secondary Outcome: Activation Profiles of NK Cells: CD16
Description: The expression levels of activation markers on NK cells profile, specifically CD16, were determined for samples collected from multiple timepoints from Week 1 to Week 70. Data is reported in the units Median Fluorescence Intensity (MFI).
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemotherapy Only arm Week 46, two participants either did not show up or were off study. For participants in Chemo+Vaccine arm Week 46 one participant either did not show up or were off study, and Week 70 three participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Median Fluorescence Intensity
  Week 1 | 72297.8 (21876.9) | 69622.91 (12067.19)
  Week 7 | 68472 (27775.62) | 72147.91 (13278.21)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 50260 (20398.6)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 56000.1 (19176)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 62015.1 (16473.61)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 66342.55 (19245.26)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 68235 (6689.29) | 57106 (26203.70)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 71401.13 (20553.46)

17. Secondary Outcome: Activation Profiles of NK Cells: CD69
Description: The expression levels of activation markers on NK cells profile, specifically CD69, were determined for samples collected from multiple timepoints from Week 1 to Week 70. Data is reported in the units Median Fluorescence Intensity (MFI).
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: Chemotherapy Only and Chemo+Vaccine arms have different schedules of activities. For participants in Chemo+Vaccine arm Week 46 one participant either did not show up or were off study, and Week 70 three participants either did not show up or were off study.
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Median Fluorescence Intensity
  Week 1 | 374.2 (19.05) | 384.1 (52.52)
  Week 7 | 396.8 (62) | 445.55 (67.32)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 423.64 (71.43)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 418.73 (54.77)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 419.82 (64.15)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 439.64 (62.75)
  Week 46: number analyzed (Participants) | 5 | 10
  Week 46 | 343 (11.5) | 413.4 (53.91)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 389.63 (79.45)

18. Secondary Outcome: Activation Profiles of NK Cells: NKp46
Description: The expression levels of activation markers on NK cells profile, specifically NKp46, were determined for samples collected from multiple timepoints from Week 1 to Week 70. Data is reported in the units Median Fluorescence Intensity (MFI).
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Median Fluorescence Intensity
  Week 1 | 997.8 (97.72) | 1206.5 (451.05)
  Week 7 | 1424.2 (592.34) | 1329.64 (578.46)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 2435.9 (1237.85)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 2600.82 (1161.2)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 2352.18 (932.15)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 1694.18 (754.75)
  Week 46: number analyzed (Participants) | 5 | 10
  Week 46 | 940.67 (221.44) | 1785.4 (664.66)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 1584.88 (452.15)

19. Secondary Outcome: Activation Profiles of NK Cells: NKG2D
Description: The expression levels of activation markers on NK cells profile, specifically NKG2D, were determined for samples collected from multiple timepoints from Week 1 to Week 70. Data is reported in the units Median Fluorescence Intensity (MFI).
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, and 70
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Median Fluorescence Intensity
  Week 1 | 900.2 (212.32) | 1050.6 (344.35)
  Week 7 | 776.2 (206.53) | 992.91 (388.52)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 1059.18 (328.94)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 1034.55 (365.92)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 941.27 (346.34)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 973.55 (283.06)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 589 (159.6) | 738.6 (142.82)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 795.38 (191.53)

20. Secondary Outcome: Activation Profiles of T Cells - CD69 on CD3+
Description: The expression levels of activation markers CD69 on T cells were determined by flow cytometry for samples collected from multiple timepoints from Week 1 to Week 70. Data is reported in the units Median Fluorescence Intensity (MFI).
Time Frame: Weeks 1, 7, 10, 15, 18, 23, 46, 70
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity (MFI)
Arm/Group | Chemotherapy Only | Chemo+Vaccine
Number analyzed (Participants) | 5 | 11
Median Fluorescence Intensity (MFI)
  Week 1 | 368.8 (31) | 394.55 (64.34)
  Week 7 | 403.2 (62.35) | 411.27 (63.6)
  Week 10: number analyzed (Participants) | 0 | 11
  Week 10 |  | 436 (86.79)
  Week 15: number analyzed (Participants) | 0 | 11
  Week 15 |  | 412.27 (154.74)
  Week 18: number analyzed (Participants) | 0 | 11
  Week 18 |  | 401.09 (102.43)
  Week 23: number analyzed (Participants) | 0 | 11
  Week 23 |  | 396.73 (54.14)
  Week 46: number analyzed (Participants) | 3 | 10
  Week 46 | 382.33 (68.12) | 388.8 (92.09)
  Week 70: number analyzed (Participants) | 0 | 8
  Week 70 |  | 333.38 (34.1)

ADVERSE EVENTS:
Time Frame: Week 1 to Week 70
Groups:
- Control Arm: Control arm: SoC neoadjuvant chemotherapy starting week 1. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Doxorubicin: Chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  Cyclophosphamide: chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG three times. Vaccine administered on weeks 1, 2 and 3 prior to chemotherapy. Subject will start their SoC neoadjuvant chemotherapy on week 4 as described above.
  Paclitaxel: chemo+vaccine arm immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4 as described above
- Chemo+Vaccine Arm: Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG three times. Vaccine administered on weeks 1, 2 and 3 prior to chemotherapy. Subjects will start their SoC neoadjuvant chemotherapy on week 4. Doxorubicin and cyclophosphamide (AC) will be administered concurrently every two weeks for four cycles with pegfilgrastim (or equivalent growth factor) on day 2 of each AC cycle, followed by paclitaxel weekly x 12 weeks.
  P10s-PADRE with MONTANIDE™ ISA 51 VG: Subjects randomized to the control arm will receive SoC neoadjuvant chemotherapy starting on week 1.
  Doxorubicin: Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4.
  Cyclophosphamide: Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4.
  Paclitaxel: Subjects randomized to the chemo+vaccine arm will be immunized with P10s-PADRE in MONTANIDE™ ISA 51 VG a total of three times. The vaccine will be administered on weeks 1, 2 and 3 prior to chemotherapy. Then, they will start their SoC neoadjuvant chemotherapy on week 4.
Arm/Group | Control Arm | Chemo+Vaccine Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/11
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/11
Other Adverse Events (participants affected / at risk) | 5/5 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=5) | Chemo+Vaccine Arm (N=11)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Vascular Disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1) — Evidence of acute deep vein thrombosis in the L mid femoral, popliteal, and posterior tibial veins
Infection and infestations, other, specify (Infections and infestations) | 0 (0) | 1 (1) — COVID 19
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=5) | Chemo+Vaccine Arm (N=11)
Anemia (Blood and lymphatic system disorders) | 5 (18) | 11 (53)
Fatigue (General disorders) | 5 (11) | 11 (47)
Lymphocyte count decreased (Investigations) | 5 (24) | 11 (104)
Investigations, Other (Investigations) | 5 (25) | 10 (60)
Nausea (Gastrointestinal disorders) | 5 (12) | 9 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (14)
White Blood Cells Decreased (Investigations) | 4 (7) | 9 (36)
Diarrhea (Gastrointestinal disorders) | 5 (8) | 7 (14)
Skin and subcutaneous disorders, other (Skin and subcutaneous tissue disorders) | 5 (9) | 7 (15)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (6) | 7 (20)
Injection Site Reaction (General disorders) | 0 (0) | 10 (21)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6) | 7 (19)
Mucositis Oral (Gastrointestinal disorders) | 3 (6) | 7 (15)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5) | 6 (14)
Depression (Psychiatric disorders) | 1 (1) | 8 (15)
Insomnia (Psychiatric disorders) | 1 (2) | 8 (13)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 7 (17)
Headache (Nervous system disorders) | 3 (5) | 5 (12)
Vomiting (Gastrointestinal disorders) | 3 (7) | 5 (11)
Hypertension (Vascular disorders) | 4 (5) | 4 (8)
Anxiety (Psychiatric disorders) | 2 (5) | 6 (8)
Alkaline Phosphatase Increased (Investigations) | 3 (7) | 4 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 7 (13)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 6 (10)
Creatinine increased (Investigations) | 1 (8) | 6 (14)
Dizziness (Nervous system disorders) | 1 (1) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7)
Breast Pain (Reproductive system and breast disorders) | 2 (2) | 5 (8)
Gastrointestinal Disorders, Other (Gastrointestinal disorders) | 2 (3) | 5 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Edema Limbs (General disorders) | 1 (1) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (5)
Pain (General disorders) | 1 (3) | 4 (10)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 4 (6)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 4 (5)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 3 (3)
Eye disorders - Other (Eye disorders) | 0 (0) | 4 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 4 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 3 (4)
Platelet count decreased (Investigations) | 1 (1) | 3 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (7)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Vascular disorder - other (Vascular disorders) | 1 (2) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Infection and infestation - other (Infections and infestations) | 0 (0) | 3 (3)
Nervous system disorders - other (Nervous system disorders) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Reproductive system and breast disorders - other (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cholesterol high (Investigations) | 0 (0) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Localized edema (General disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiac Disorders - other (Cardiac disorders) | 0 (0) | 1 (2)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
GGT increased (Investigations) | 0 (0) | 1 (3)
INR increased (Investigations) | 0 (0) | 1 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Nail Loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (2) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Social circumstances - other (Social circumstances) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT02938442/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02938442/ICF_002.pdf